CLINICAL TRIAL: NCT00509873
Title: A Study of the Safety and Efficacy of Gatifloxacin in Patients With Bacterial Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 198782-004
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-10

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Gatifloxacin; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Gatifloxacin 0.5% Eye Drops (Experimental): Gatifloxacin 0.5% Eye Drops
  Interventions: Drug: Gatifloxacin 0.5% eye drops
- Placebo Eye Drops (Placebo Comparator): Placebo Eye Drops
  Interventions: Drug: placebo eye drops

INTERVENTIONS:
Drug: Gatifloxacin 0.5% eye drops — Day 1 = 1 drop of study medication every 2hrs up to 8 times total; day 2-5 = 1 drop twice daily
  Arms: Gatifloxacin 0.5% Eye Drops
Drug: placebo eye drops — Day 1 = 1 drop of study medication every 2hrs up to 8 times total; day 2-5 = 1 drop twice daily
  Arms: Placebo Eye Drops

SUMMARY:
The study will determine the safety and efficacy of gatifloxacin eye drops in patients with bacterial conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with bacterial conjunctivitis

Exclusion Criteria:

* Signs and/or symptoms of conjunctivitis for more than 96 hours
* Signs and/or symptoms suggestive of fungal, viral, or allergic conjunctivitis
* Clinical diagnosis of chlamydia in either eye

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Gretna, Louisiana, United States

REFERENCES:
- [Derived] Heller W, Cruz M, Bhagat YR, De Leon JM, Felix C, Villanueva L, Hollander DA, Jensen H. Gatifloxacin 0.5% administered twice daily for the treatment of acute bacterial conjunctivitis in patients one year of age or older. J Ocul Pharmacol Ther. 2014 Dec;30(10):815-22. doi: 10.1089/jop.2014.0040. PMID 25244402

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Started | 287 | 291
Completed | 276 | 276
Not Completed | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops | Total
Number analyzed (Participants) | 287 | 291 | 578
Age, Customized [Number; unit: participants]
  1-18 years | 123 | 123 | 246
  19-65 years | 126 | 141 | 267
  >65 years | 38 | 27 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 172 | 333
  Male | 126 | 119 | 245

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Clearing (Clinical Success) of Conjunctival Hyperemia and Conjunctival Discharge at Day 6
Description: Percentage of patients that achieved clinical success, defined as achievement of a score of zero for both conjunctival hyperemia and conjunctival discharge in the study eye at Day 6. Conjunctival hyperemia and conjunctival discharge were each assessed on a 4-point severity grade scale (0=none, +1=mild, +2=moderate, +3=severe).
Time Frame: Day 6
Population: Modified Intent to Treat; defined as all randomized patients who were "culture positive" at baseline meaning the culture of the eye grew bacteria. (Note: The Day 6 analysis included all Day 6 visit data, regardless of whether it was collected on Day 6 or on a later day).
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 167 | 158
Percentage of Patients | 74.9 | 65.2

2. Secondary Outcome: Percentage of Patients With Microbiological Cure at Day 6
Description: Percentage of patients with microbiological cure, defined such that all bacteria present in the study eye at Day 1 (Baseline) are eradicated (or absent) at Day 6 based on a Classification of Microbial Response. (Eradication=pathogen is absent in follow-up culture; Reduction=pathogen is reduced from baseline below threshold count in follow-up culture; Persistence=pathogen reduced from baseline but is above or equal to threshold count in follow-up culture; and Proliferation=pathogen has increased in count from baseline in follow-up culture)
Time Frame: Day 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 167 | 158
Percentage of Patients | 89.2 | 61.4

3. Secondary Outcome: Percentage of Patients With Clinical Improvement of Ocular Signs at Day 6
Description: Percentage of patients with clinical improvement of ocular signs at Day 6 based on a 4-point scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe), defined as a decrease (improvement) from Day 1 (Baseline) in the total score of conjunctival hyperemia and mucopurulent discharge (pus),with no increase (worsening) from Day 1 (Baseline) in either individual variable in the study eye.
Time Frame: Day 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 167 | 158
Percentage of Patients | 97.0 | 96.2

4. Secondary Outcome: Percentage of Patients With Clinical Improvement of Ocular Symptoms at Day 6
Description: Percentage of patients with clinical improvement of ocular symptoms at Day 6, defined as a decrease (improvement) from Day 1 (Baseline) in the total score of itching and tearing (each on 4-point scale: 0 = none, 1 = mild, 2 = moderate, and 3 = severe), with no increase (worsening) from Day 1 (Baseline) in any individual score in the study eye diagnosed with bacterial conjunctivitis
Time Frame: Day 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 167 | 158
Percentage of Patients | 85.5 | 82.2

5. Post Hoc Outcome: Percentage of Patients With Clearing (Clinical Success) of Conjunctival Hyperemia and Conjunctival Discharge Up to Day 6
Description: Percentage of patients that achieved clinical success, defined as achievement of a score of zero for both conjunctival hyperemia and conjunctival discharge in the study eye up to Day 6. Conjunctival hyperemia and conjunctival discharge were each assessed on a 4-point severity grade scale (0=none, +1=mild, +2=moderate, +3=severe). (Note: The "Up to Day 6" analysis included all data up to the Day 6 time point but excluded any Day 6 visit data that was collected after the Day 6 time point).
Time Frame: 6 Days
Population: Modified Intent to Treat; defined as all randomized patients who were "culture positive" at baseline meaning the culture of the eye grew bacteria. (Note: The "Up to Day 6" analysis included all data up to the Day 6 time point but excluded any Day 6 visit data that was collected after the Day 6 time point).
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 167 | 158
Percentage of Patients | 64.1 | 50.0

ADVERSE EVENTS:
Description: Safety Population used for serious adverse event and adverse event analysis - defined as all patients who were randomized AND treated based on actual treatment received.
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Serious Adverse Events (participants affected / at risk) | 0/288 | 1/289
Other Adverse Events (participants affected / at risk) | 14/288 | 13/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gatifloxacin 0.5% Eye Drops (N=288) | Placebo Eye Drops (N=289)
Cardiac failure congestive (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gatifloxacin 0.5% Eye Drops (N=288) | Placebo Eye Drops (N=289)
Conjunctivitis bacterial (Infections and infestations) | 14 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.